CLINICAL TRIAL: NCT06181097
Title: Routine Use of Negative Pressure Wound Therapy in Primary Hip and Knee Arthroplasties; a Randomized Controlled Trial
Brief Title: Routine Use of Negative Pressure Wound Therapy THR TKR RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Tim-Yun Michael ONG, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.208
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Knee Arthropathy; Hip Arthropathy; Negative Pressure Wound Therapy
Keywords: Knee Arthropathy; Hip Arthropathy; TKR; THR; Wound therapy
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: Eligible patients will be recruited and randomized to either NPWT and standard dressing.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- negative pressure wound therapy (Experimental): Both groups will have layered closure with 2-O Vicryl (polyglactin 910) braided suture for the subcutaneous layers and 3-O Stratafix knotless barbed suture for the subcuticular layer. Fixation strips (STERI-Strip, 3M) would then be applied to the entire length of the wound. For the NPWT group, the Smith & Nephew PICO dressing will be chosen as it is versatile with various size options, and the small suction pump is would not causing much problems to patient mobility. For the standard dressing group, the same PICO dressing will be applied, but without the suction.
  Interventions: Device: negative pressure wound therapy
- standard dressing (Active Comparator): Both groups will have layered closure with 2-O Vicryl (polyglactin 910) braided suture for the subcutaneous layers and 3-O Stratafix knotless barbed suture for the subcuticular layer. Fixation strips (STERI-Strip, 3M) would then be applied to the entire length of the wound. For the NPWT group, the Smith & Nephew PICO dressing will be chosen as it is versatile with various size options, and the small suction pump is would not causing much problems to patient mobility. For the standard dressing group, the same PICO dressing will be applied, but without the suction.
  Interventions: Other: standard dressing

INTERVENTIONS:
Device: negative pressure wound therapy — The intervention group will have layered closure with a 2-O Vicryl (polyglactin 910) braided suture for the subcutaneous layers and a 3-O Stratafix knotless barbed suture for the subcuticular layer. Fixation strips (STERI-Strip, 3M) would then be applied to the entire length of the wound. The Smith & Nephew PICO dressing will be chosen as it is versatile with various size options, and the small suction pump is would not causing much problems to patient mobility.
  Arms: negative pressure wound therapy
Other: standard dressing — The standard dressing group will have layered closure with a 2-O Vicryl (polyglactin 910) braided suture for the subcutaneous layers and a 3-O Stratafix knotless barbed suture for the subcuticular layer. Fixation strips (STERI-Strip, 3M) would then be applied to the entire length of the wound. The same PICO dressing will be applied, but without the suction.
  Arms: standard dressing

SUMMARY:
Negative pressure wound therapy (NPWT) for post total joint arthroplasty incisions has demonstrated benefits in reducing wound complications. A prospective randomized trial will be conducted including 40 patients who will undergo total knee and total hip arthroplasty. The number of wound complications within 21 days will be recorded. As well, the aesthetic appearance and quality of scarring of the scar will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total knee or total hip arthroplasty at Prince of Wales Hospital, Hong Kong.

Exclusion Criteria:

* Patients using steroid, or other immune modulators that is known to affect wound healing, prior surgery to the knee or hip, skin condition such as eczema that would result in poor healing or widen scars, patients with a known significant history of hypertrophic scarring or keloid.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Wound-related complications | 21 days after surgery
  Recurrence of wound exudate, surgical site infections, dressing-related issues, readmission to hospital and any further surgical interventions will be documented by the research personnel status at 21 days after the index operation.

SECONDARY OUTCOMES:
Patient Scale and Observer Scale (POSAS) | 21 days after surgery
  The POSAS has category boxes to core nominal parameters, for example colour of the scar. Each item of both scales have a 10-point score, with 10 indicating the worse imaginable scar or sensation and 1 corresponding to normal scar or skin (normal pigmentation, no itching, etc.). The total score of both scale is calculated by summing up the score of each of the six items and ranges from 6 to 60.
Multi-category visual analogue scale | 21 days after surgery
  The multi-category visual analogue scale (VAS) is a photograph based scale derived from evaluating standardised digital photographs in four categories (pigmentation, vascularity, acceptability and patient comfort) plus contour. The individual scores are added to give a single overall score ranging from "excellent" to "poor"

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: Journal reviewers